CLINICAL TRIAL: NCT01343836
Title: The Value of Autologous Tenocyte Implantation in Patients With Chronic Achilles Tendinopathy: a Double-blind Randomised Clinical Trial
Brief Title: Autologous Tenocyte Implantation in Patients With Chronic Achilles Tendinopathy
Acronym: ATI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Prof J.A.N. Verhaar, Prof. J.A.N. Verhaar, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: METC10-102
Record Dates: First submitted 2011-04-27; First posted 2011-04-28 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Tendinopathy; Achilles Tendon Injury; Achillodynia
Keywords: autologous tenocytes; cell therapy; eccentric exercises
MeSH Terms: conditions — Tendinopathy | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Autologous Tenocyte Implantation (Experimental): Intratendinous ATI (autologous tenocyte implantation) injection with eccentric exercises
  Interventions: Other: Autologous Tenocyte Implantation
- Saline injection (Placebo Comparator): Intratendinous saline injection with eccentric exercises
  Interventions: Other: Saline

INTERVENTIONS:
Other: Autologous Tenocyte Implantation — Intratendinous ATI (autologous tenocyte injection) with eccentric exercises
  Arms: Autologous Tenocyte Implantation
Other: Saline — Intratendinous saline injection with eccentric exercises
  Arms: Saline injection

SUMMARY:
This study is designed to compare the treatment of 2 groups in patients with Achilles tendinopathy: autologous tenocytes injection in combination with exercises versus saline injection in combination with exercises

DETAILED DESCRIPTION:
Overuse injury of the Achilles tendon is a common entity. When the exact origin of tendon pain is unclear, the term tendinopathy is preferred. Most accepted treatment at this moment is an eccentric exercise programme, according to the Dutch guidelines. However, a recent systematic review on the effectiveness of eccentric exercises to treat lower extremity tendinoses concluded that it is unclear whether eccentric exercises are more effective than other forms of treatment. Recent studies described new treatment strategies in tendinopathies, such as the use autologous Tenocyte Implantation (ATI). This treatment option can participate actively in tissue repair processes on cell level. The only published clinical pilot study in tendon research reported 60% improvement in all scores after 6 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Pain on palpation 2-7 cm proximal from the tendon insertion ("midportion")
* Symptoms > 2 months
* Age 18-55 years

Exclusion Criteria:

* Clinical suspicion of insertional disorders , Achilles tendon rupture, plantar flexor tenosynovitis, sural nerve pathology, peroneal subluxation
* Condition of the Achilles tendon caused by medications such as quinolones and statins
* Known to have the following disorders: spondylarthropathy, gout, hyperlipidemia, rheumatoid arthritis and sarcoidosis.
* Antibiotics allergy (aminoglycoside group)
* A condition that prevents the patients from executing an active rehabilitation programme
* Patient has received an injection for this injury
* Patient has received surgical intervention for this injury
* Patient has already one site (left or right) included in this study
* Patient does not wish, for whatever reason, to undergo one of the two treatments
* Known pregnancy
* Nursing women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2011-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
VISA-A score | 24 weeks
  a validated instrument to detect the severity of symptoms in patients with Achilles tendinopathy

SECONDARY OUTCOMES:
Ultrasonographic tendon repair - Ultrasonographic Tissue Characterization (UTC) | 24 weeks
  UTC provides quantitative information on tendon fiber alignment and the related ultra-structural integrity of the tendon tissue through a non-invasive approach and is used in several clinical trials in humans
Subjective patient satisfaction | 24 weeks
  Patient satisfaction will be determined by asking the patient how satisfied he/she is with the effect of the treatment in 4 possible categories: excellent / good / moderate / poor. The groups "excellent" and "good" will be regarded as successful and the groups of "moderate" and "poor" as not successful.
Returning to sports level | 24 weeks
  The patient will be asked whether they are able to return to their sports level. It is a subdivision in 5 groups: A. No sports; B. No return in sports; C. Returning in sports but not in desired sport; D. Returning in desired sport, but not yet old level; E. Returning to old level in desired sport.

CONTACTS AND LOCATIONS:
Overall Officials: J.A.N. Verhaar, Prof, Principal Investigator — Erasmus Medical Center; P.L.J. van Veldhoven, MD, Principal Investigator — Medical Center The Hague
Locations (1):
- Sports medicine department Medical Center The Hague, Leidschendam, South Holland, Netherlands

REFERENCES:
- [Background] Chen J, Yu Q, Wu B, Lin Z, Pavlos NJ, Xu J, Ouyang H, Wang A, Zheng MH. Autologous tenocyte therapy for experimental Achilles tendinopathy in a rabbit model. Tissue Eng Part A. 2011 Aug;17(15-16):2037-48. doi: 10.1089/ten.TEA.2010.0492. Epub 2011 Jun 10. PMID 21495863